CLINICAL TRIAL: NCT05891483
Title: A Multicentre, Randomised, Double-Blind, Placebo-Controlled, Parallel-Group Phase 2 Efficacy and Safety Study of SHR-1905 in Patiens With Chronic Rhinosinusitis With Nasal Polyps
Brief Title: Efficacy and Safety of SHR-1905 Injection in Patients With Chronic Rhinosinusitis With Nasal Polyps
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1905-202
Record Dates: First submitted 2023-05-25; First posted 2023-06-07 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group A: SHR-1905 Injection（dose 1） (Experimental)
  Interventions: Drug: SHR-1905 Injection
- Treatment group B: SHR-1905 Injection（dose 2） (Experimental)
  Interventions: Drug: SHR-1905 Injection
- Treatment group C: SHR-1905 Injection（dose 3） (Experimental)
  Interventions: Drug: SHR-1905 Injection
- Placebo Group (Placebo Comparator)
  Interventions: Drug: SHR-1905 Placebo Injection

INTERVENTIONS:
Drug: SHR-1905 Injection — SHR-1905 Injection
  Arms: Treatment group A: SHR-1905 Injection（dose 1）; Treatment group B: SHR-1905 Injection（dose 2）; Treatment group C: SHR-1905 Injection（dose 3）
Drug: SHR-1905 Placebo Injection — SHR-1905 Placebo Injection
  Arms: Placebo Group

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of SHR-1905 injection in subjects with chronic rhinosinusitis with nasal polyps (CRSwNP), as well as to explore the reasonable dosage of SHR-1905 injection for CRSwNP.

ELIGIBILITY:
Inclusion Criteria:

1. Weight ≥40kg
2. Diagnosed with chronic rhinosinusitis with nasal polyps (CRSwNP).
3. Bilateral nasal polyps at screening and baseline, total NPS ≥5, ≥2 points for each nostril.
4. NCS ≥2 at screening and baseline.
5. SNOT-22≥20 at screening period and baseline.
6. Recorded persistent NP symptoms for over 4 weeks prior to screening.
7. Subjects received standard therapy with intranasal corticosteroids (INCS) and remained stable during the 4 weeks prior to randomization.
8. NP surgery in the past and/or ACERS treated with SCS occurred within 2 years before randomization (or with contraindications/ intolerances).

Exclusion Criteria:

1. Any comorbidities that may affect the efficacy evaluation of nasal polyps.
2. Any comorbidities except for asthma that may affect blood EOS levels.
3. Concomitant with immunodeficiency.
4. Concomitant with contraindications or not suitable for nasal endoscopy.
5. Uncontrolled hypertension.
6. Uncontrolled diabetes.
7. Infection within 2 weeks prior to screening to randomization that is clinically significant and/or should be treated with systemic antibiotics.
8. Uncontrolled epistaxis within 4 weeks prior to randomization.
9. Major surgery performed within 3 months prior to randomization, or surgery planned during the study, or treatments that may affect evaluations according to investigators.
10. Parasitic infection within 6 months before randomization.
11. Sinus or intranasal surgery (except for diagnostic biopsy) within 6 months prior to randomization, or changes in the nasal walls caused by sinus or intranasal surgery that made NPS evaluation impossible.
12. Malignancies diagnosed within 5 years before randomization (except those with a low risk of metastasis or death).
13. Abnormalities of laboratory tests at screening or baseline.
14. Concomitant with active hepatitis B, positive hepatitis C virus antibodies, positive human immunodeficiency virus antibodies, or positive treponema pallidum antibodies.
15. Prolonged QTc interval (>450ms for male and >470ms for female) or other clinically significant abnormal results of ECG at screening or baseline that may cause significant safety risks to subjects.
16. FEV1 before the use of bronchodilator (pre-BD) was less than 50% at screening.
17. Transfusion of blood products or immunoglobulin within 4 weeks prior to randomization.
18. SCS or additional INCS use within 4 weeks before randomization, or planned use during treatment period.
19. Regular use of decongestants (local or systemic) within 4 weeks before randomization, except for during the endoscopic procedure.
20. Adnimistration of live vaccine or viral vector vaccine within 4 weeks before randomization.
21. Allergen immunotherapy within 8 weeks before randomization.
22. Smoking history ≥10 pack-years, smoking at screening, or smoking cessation less than 6 months at screening.
23. Substance abuse, drug abuse, and/or excessive alcohol consumption within 1 year prior to randomization.
24. Pregnancy (including positive pregnancy test at screening or baseline), lactation, or pregnancy plan during study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Nasal polyp scores (NPS) | Baseline to Week 24
  Change from baseline in NPS at Week 24.

SECONDARY OUTCOMES:
NPS | Baseline to Week 48
  Changes from baseline in NPS from baseline at each evaluation time point.
Nasal Congestion Scores (NCS) | Baseline to Week 48
  Changes from baseline in NCS at each evaluation time point.
Loss of smell | Baseline to Week 48
  Changes from baseline in scores of loss of smell at each evaluation time point.
Runny nose/postnasal drip | Baseline to Week 48
  Change from baseline in scores of runny nose/postnasal drip at each evaluation time point.
Facial pain and/or pressure | Baseline to Week 48
  Change from baseline in facial pain and/or pressure scores at each evaluation time point.
Total symptoms score (TSS) | Baseline to Week 48
  Changes from baseline in TSS each evaluation time point.
Sino-nasal outcome test-22 (SNOT-22) scores | Baseline to Week 48
  Changes from baseline in SNOT-22 scores at each evaluation time point.
Proportion of subjects exposed to SCS for acute exacerbation of chronic rhinosinusitis (AECRS) over 24 weeks. | Baseline to Week 24
Dose of SCS used for AECRS over 24 weeks (converted to equivalent dose of prednisone). | Baseline to Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & Ent Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided